CLINICAL TRIAL: NCT07220941
Title: Efficacy and Feasibility of an Online Acceptance Based Intervention for Misophonia: A Randomized Controlled Trial
Brief Title: Digital Intervention for Adults With Misophonia: A Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Utah State University (Other)
Collaborators: Misophonia Research Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15239
Record Dates: First submitted 2025-10-21; First posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Misophonia
Keywords: Acceptance and commitment therapy (ACT); Digital mental health intervention (DMHI)
MeSH Terms: conditions — misophonia | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT online program (Experimental): Participants will complete the 8-module fully automated digital intervention based in acceptance and commitment therapy (ACT).
  Interventions: Behavioral: Acceptance and commitment therapy
- Waitlist Control (No Intervention): Waitlist condition; assessment only.

INTERVENTIONS:
Behavioral: Acceptance and commitment therapy — Participants will complete the 8-module fully automated digital intervention based in acceptance and commitment therapy (ACT). The digital program is based off of an ACT protocol developed in a prior randomized controlled trial and adapted for digital self-help use (Bowers et al., 2024). Modules focus on focus on acceptance, cognitive defusion, present moment awareness, values clarification, and functional adaptations.
  Other Names: ACT
  Arms: ACT online program

SUMMARY:
The goal of this clinical trial is to test an online intervention for adults with misophonia. The main questions it aims to answer are:

1. Is the online intervention effective, compared to a waitlist control condition?
2. Is the online intervention acceptable to use?

Participants will be randomized into either the online intervention or waitlist control condition:

1. Participants in the intervention condition will be asked to complete an 8 module acceptance and commitment therapy (ACT) program for misophonia and 5 surveys over 4 months.
2. Participants in the waitlist condition will be asked to complete 5 surveys over 4 months, and will receive access to the intervention once the study is complete.

DETAILED DESCRIPTION:
Misophonia, characterized by intense emotional reactions to specific sounds, significantly impacts daily functioning and quality of life. Acceptance and Commitment Therapy (ACT) has shown promise in addressing misophonia symptoms by fostering psychological flexibility. While recent intervention studies demonstrate the efficacy of ACT for misophonia, accessible and scalable treatment options remain scarce. This study aims to address this gap by developing and evaluating a fully automated, online ACT-based digital mental health intervention for misophonia. We will compare the intervention to a delayed treatment group in a sample of 100 adults meeting clinical criteria for misophonia. Outcomes will include misophonia symptoms, quality of life, general distress, and psychological flexibility, assessed at baseline, mid-intervention, post-intervention, and one- and two-month follow-up. Multilevel modeling will test time by condition interactions to examine the efficacy and feasibility of an online ACT-based intervention. This fully automated online intervention aims to provide accessible, evidence-based treatment for individuals with misophonia, laying groundwork for future, larger-scale studies and public dissemination.

ELIGIBILITY:
Inclusion Criteria:

* Currently meet clinical impairment for misophonia.
* At least 18 years old.
* Fluent English speakers.
* Currently live or reside in the United States

Exclusion Criteria:

* Currently receiving alternative psychotherapy for misophonia.
* Currently modifying or starting psychotropic medication (within 30 days of starting the study).
* Any psychological and/or neurological impairments that would preclude someone from participating in the study (e.g.,active self-harm or psychosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Selective Sound Sensitivity Syndrome Scale (S-Five; Vitoratou et al., 2021) | 16 weeks
  The S-Five is a 25-item self-report measure of misophonia severity. Items (e.g., "I feel trapped if I cannot get away from certain noises") are rated on a 0 (not at all true) to 10 (completely true) ordinal scale with total scores ranging from 0 to 250. The S-Five consists of five latent factors: (1) externalizing appraisals (e.g., blaming others for making sounds), (2) internalizing appraisals (e.g., negative self-judgments triggered by misophonia), (3) impact on functioning (e.g., social and occupational impact), (4) outburst (e.g., experiences of aggression or fear of losing control), and (5) threat (e.g., feeling trapped or helpless). The S-Five demonstrates good internal consistency and convergent validity with other misophonia measures (Vitoratou et al., 2023).

SECONDARY OUTCOMES:
Misophonia acceptance and action questionnaire (Miso-AAQ; Capel et al., 2025) | 16 weeks
  The Miso-AAQ is a 7-item self-report measure of misophonia-specific psychological inflexibility, adapted from the AAQ-III (Ong et al., 2019). Items (e.g., "I'm so afraid of my reactions to sounds that I don't do things I care about" are rated from 1 (never true) to 7 (always true) Likert scale. Total scores range from 7 to 49 with higher scores indicating greater misophonia-specific psychological inflexibility. Preliminary validation from a treatment seeking sample of adults with misophonia suggest good internal consistency and convergent validity (Capel et al., 2025).
Comprehensive assessment of Acceptance and Commitment Therapy processes (CompACT; Francis et al., 2016) | 16 weeks
  The CompACT is a 23-item self-report measure of psychological flexibility. Items (e.g., "I make choices based on what is important to me, even if it is stressful) are rated on a 7-point Likert scale from 0 (strongly disagree) to 6 (strongly agree), with 12 items reverse-scored. Total scores range from 0 to 138 with higher scores indicating greater psychological flexibility. The CompACT demonstrates good internal consistency and convergent validity (Francis et al., 2016).
Depression Anxiety Stress Scale (DASS-21; Lovibond & Lovibond, 1995) | 16 weeks
  The DASS-21 is a 21 item self-report measure of distress comprised of three 7-item subscales: (1) depression, (2) anxiety, and (3) stress. Items are rated from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time), with higher scores indicating greater symptom severity. Subscale scores are summed and multiplied by two, yielding scores ranging from 0-42 for each subscale.
Mental Health Continuum-Short Form (MHC-SF; Keyes, 2005) | 16 weeks
  The MHC-SF is a 14-item self-report measure of well-being. Items assess emotional, social, and psychological well-being, rated on a 6-point Likert scale from 0 (never) to 5 (every day). A total score is calculated from summing all items and ranges from 0 to 70, with higher scores reflecting greater well-being. The MHC-SF has demonstrated strong internal consistency and validity in prior studies (Lamers et al., 2011).

OTHER OUTCOMES:
Internalized Health-Related Stigma Scale (I-HEARTS; Pearl et al., 2024) | 16 weeks
  The I-HEARTS is a 25-item self-report measure assessing internalized health-related stigma, adapted here to reference misophonia specifically. Items (e.g., "I am embarrassed or ashamed that I have misophonia") are rated on a 1 (strongly disagree) to 7 (strongly agree) Likert scale, with higher scores indicating greater internalized stigma. The scale yields a total score and three subscales: (1) perceived and anticipated stigma, (2) stereotype application and self-devaluation, and (3) stigma resistance (reverse-scored). Validation in a large sample of adults with chronic health conditions demonstrated strong internal consistency, test-retest reliability, and convergent validity with related constructs such as shame, loneliness, and depression (Pearl et al., 2024).
Interpersonal Reactivity Index - Perspective Taking (IRI-PT; Davis, 1980) | 16 weeks
  The IRI-PT is a 7-item self-report subscale assessing the tendency to adopt others' psychological perspectives. Items (e.g., "Before criticizing somebody, I try to imagine how I would feel if I were in their place") are rated from 0 (does not describe me well) to 4 (describes me very well). Total scores range from 0 to 28, with higher scores indicating greater perspective-taking propensity. The IRI-PT has demonstrated good internal consistency and validity as a measure of perspective taking (Davis, 1980).

CONTACTS AND LOCATIONS:
Overall Officials: Emily M Bowers, M.S., Principal Investigator — Utah State University
Locations (1):
- Utah State University, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: No